CLINICAL TRIAL: NCT00509015
Title: Mass-Drug Administration With a Gametocytocidal Drug Combination, a Model for a Transmission Blocking Vaccine
Brief Title: Mass-Drug Administration to Reduce Malaria Transmission
Acronym: MDATRANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Seif Shekalaghe, Kilimanjaro Christian Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APRIORI1/01
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Malaria, Falciparum
Keywords: antimalarials; malaria transmission; mass drug administration; artemisinin-based combination therapy; primaquine; gametocytes; QT-NASBA
MeSH Terms: conditions — Malaria, Falciparum | interventions — fanasil, pyrimethamine drug combination; Artesunate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Sulphadoxine-pyrimethemine (day 1) artesunate (day 1-3) primaquine (day 3)
  Interventions: Drug: Sulphadoxine-pyrimethamine (day 1: 500mg S&25mg P/20 kg); Drug: Artesunate (day 1,2,3: 4 mg/kg); Drug: Primaquine-base (day 3: 0.75 mg/kg)
- 2 (Placebo Comparator): Placebo: lactose tablets (Albochin)
  Interventions: Drug: placebo tablets

INTERVENTIONS:
Drug: Sulphadoxine-pyrimethamine (day 1: 500mg S&25mg P/20 kg) — 500mg S&25mg P/20 kg, 1 day, single dose
  Arms: 1
Drug: Artesunate (day 1,2,3: 4 mg/kg) — 4 mg/kg, daily single dose over three days
  Arms: 1
Drug: Primaquine-base (day 3: 0.75 mg/kg) — single dose at 0.75 mg/kg on day 3
  Arms: 1
Drug: placebo tablets — 3 days of lactose tablets (160mg) albochin
  Arms: 2

SUMMARY:
In the 1950s, the WHO included mass drug administration (MDA) with antimalarial drugs as a tool for malaria control in 'exceptional conditions when conventional control strategies have failed'. Subsequently, MDA has received little attention until the introduction of artemisinin based combination therapy (ACT). The principle aim of MDA is to interrupt malaria transmission by clearing the population of sexual stage parasites, gametocytes, prior to the transmission season. Gametocytes are essential for propagation of the disease and elimination of gametocytes will result in a reduction in malaria transmission. As a consequence, a successful MDA will reduce the burden of disease in a population and is expected to have little influence on the development of protective immunity in areas of low transmission intensity. In Africa, only one large scale MDA study was conducted in the last 10 years. That study, conducted in The Gambia using sulphadoxine-pyrimethamine (SP) plus a single dose of artesunate (AS), failed to show a significant impact of MDA on malaria transmission. Possible reasons for this failure are the limited impact of the drug regimen (a single dose of AS) on malaria transmission, the incomplete coverage, the relatively high transmission intensity in the area and the migration of individuals between villages. Here, we propose to conduct an MDA study in an area of very low malaria transmission intensity in Tanzania. We use the highly active drug combination SP+AS (3 days) followed by a single dose of primaquine..

DETAILED DESCRIPTION:
1. INTRODUCTION

1.1 Mass drug administration as a public health tool In the 1950s, the WHO included mass drug administration (MDA) with antimalarial drugs as a tool for malaria control in 'exceptional conditions when conventional control strategies have failed'. Subsequently, MDA has received little attention until the introduction of artemisinin based combination therapy (ACT). The principle aim of MDA is to interrupt malaria transmission by clearing the population of sexual stage parasites, gametocytes, prior to the transmission season (figure 1). Gametocytes are essential for propagation of the disease and elimination of gametocytes will result in a reduction in malaria transmission. As a consequence, a successful MDA will reduce the burden of disease in a population and is expected to have little influence on the development of protective immunity in areas of low transmission intensity. In Africa, only one large scale MDA study was conducted in the last 10 years. That study, conducted in The Gambia using sulphadoxine-pyrimethamine (SP) plus a single dose of artesunate (AS), failed to show a significant impact of MDA on malaria transmission.1 Possible reasons for this failure are the limited impact of the drug regimen (a single dose of AS) on malaria transmission, the incomplete coverage, the relatively high transmission intensity in the area and the migration of individuals between villages. Here, we propose to conduct an MDA study in an area of very low malaria transmission intensity in Tanzania.

1.2 Drug-combinations for MDA Antimalarial drugs are only suitable for MDA if they are safe, effective in clearing asexual parasites and have a profound effect on gametocytes. Artemisinin based combination therapy fulfils all these criteria. The combination of sulphadoxine-pyrimethamine (SP) and a three dose regimen of artesunate (AS) has been extensively tested in Tanzania, Uganda and Kenya, is safe and efficacious in clearing asexual parasites and reduces gametocytaemia. In pregnant women, no negative effects of AS were reported.

SP + AS is, however, not capable of clearing all gametocytes and is therefore unable to fully prevent malaria transmission. Primaquine (PQ) is the only drug that has been shown to actively clear gametocytes.

PQ has previously been used for treating symptomatic patients in the lower Moshi area, the area where the current study will be carried out. The rationale was to reduce post-treatment malaria transmission. The strategy was abandoned to follow national guidelines but no side effects were reported. In addition, PQ was recently used in combination with SP and AS and found to be safe and highly efficacious in clearing all parasite stages. However, there is concern for negative haemolytic side effects that have been reported for the full dose regimen in individuals who are G6PD deficient. Haemolytic side effects are generally self-limiting and, more importantly, are observed in individuals receiving the full dose PQ treatment (0.5 mg/kg, 14 days). Despite these limitations of PQ as full-dose treatment, PQ can also be used to clear gametocytes, after clearing asexual parasites with a different drug or drug-combination. This gametocytocidal treatment requires a single dose of PQ only and is mentioned by the World Health Organization (WHO) as beneficial in areas of low malaria transmission. PQ has a short half-life of 5-6 hours and the single dose of 0.75mg/kg (adults 45mg) is too low to cause haemolytic effects. According to WHO standards, testing for G6PD deficiency is therefore not required.

For this study, we propose to use the standard dose of SP + AS to clear asexual parasites, followed by a single dose of PQ to clear remaining gametocytes. Pregnant women and children under 1 years of age will be excluded from PQ treatment. Prior to the proposed study, a small scale clinical study was conducted in symptomatic children in Korogwe to determine the safety and gametocytocidal effect of SP + AS and SP + AS followed by PQ (NIMR/HQ/R.8a Vol. XIII/446; http://www.controlled-trials.com/ISRCTN61534963). We did do screen for G6PD deficiency prior to treatment in this pilot study and did not observe any side effects or clinical indication of anaemia in children treated with PQ.

1.3 MDA and transmission blocking vaccines Apart from the direct benefit of MDA as a malaria control tool, the proposed study has a scientific objective to determine the suitability of several evaluation tools for a transmission blocking vaccine (TBV). TBV work by inducing antibodies that react with parasite surface antigens in the mosquito midgut after a blood meal. These immune responses suppress the infectivity to mosquitoes and can therefore potentially prevent transmission. Although several groups work on the production of a TBV, there is no experience with the evaluation of such a vaccine in the field. The evaluation of a TBV is rather different of the evaluation of a conventional vaccine which protects the vaccinated individual directly. A TBV doesn't protect the vaccinated individual but the community and has therefore to be evaluated on the community level. Limited available data regarding the protection of communities comes from studies on insecticide treated bed nets.

A successful MDA with gametocytocidal drugs could serve as a proof of principle for a transmission blocking vaccine. A MDA study is expected to have a similar impact on malaria transmission as a TBV: while the contact between man and mosquito is not influenced, the infectiousness of the human population to mosquitoes is reduced. Because of this similarity, both need identical evaluation tools. An MDA can therefore be used to test the sensitivity and suitability of clinical and biological measures.

2. OBJECTIVES

1. To determine the impact of mass drug administration with a gametocytocidal drug combination on

   1. malaria morbidity
   2. parasite prevalence
   3. the human infectious reservoir
2. To determine the suitability of outcome measures for detecting reductions in malaria transmission
3. To model the impact of MDA on malaria transmission.

3. WORK PLAN

3.1 Study area The proposed study area is an area in Lower Moshi that has been part of ongoing activities of the Kilimanjaro Christian Medical Centre/Joint Malaria Programme in since 2002 The study area is characterised by a very low transmission intensity with an entomologic inoculation rate (EIR) of 3.4 (95% CI 0.7 - 9.9) infectious bites per person per year. Despite low transmission intensity, an estimated 300-400 clinical malaria cases occur yearly, predominantly in the transmission season. In the area, 4 isolated villages were selected, mapped and censused. Malaria transmission in the villages was characterised by weekly mosquito catches and two cross-sectional surveys for parasitological parameters. Villages are comparable in entomologic and parasitological characteristics and parasite carriage as determined by microscopy (1-3%) and molecular detection techniques (30-40%) is equally distributed over different age groups (NIMR/HQ/Vol.IX/343). Two health facilities exist in the study area, both serving three villages. The health facilities are participating in passive case detection since February 2006. For the proposed study, clusters have been defined using a completed map of the study area where the coordinates of each individual house was mapped using geographical positioning system (GPS). The minimum distance between clusters is 1 kilometer. MDA with the gametocytocidal drug combination will be undertaken in approximately 8 clusters, MDA with a placebo in the other clusters. Migration in the study area will be carefully monitored by community workers. Balozi's will be actively involved in this part of the study. During a cross-sectional study that was carried out in the preparation phase of this study >98% of the individuals indicated that they were permanent residents of the area and to sleep in their house every night of the year. Possible migration of individuals during the follow-up period will be included in determining the minimum coverage of the MDA.

3.2 Intervention by mass drug administration Prior to the transmission season, all individuals will receive either mass drug administration (MDA) or placebo. This administration is done irrespective of the presence of parasites or symptoms. Treatment dosage is sulphadoxine- pyrimethamine (Fansidar, Roche, Switzerland: S 500mg/20kg; P 25mg/20kg, day1), artesunate (Arsumax, Sanofi, France: 4mg/kg, day1,2,3) and primaquine (PQ base, Radboud University Nijmegen, The Netherlands: 0.75 mg/kg) Pregnant women and children below 1 year of age will be excluded from PQ treatment.

3.3 Evaluation of the intervention Primary outcome measures for follow-up are i)malaria morbidity, ii) asexual parasite and gametocyte prevalence, iii) entomologic inoculation rate, iv) the human infectious reservoir. These measures will be determined on several occasions over 6 months.

i) Malaria morbidity is assessed by passive case detection in two health centres and by active case detection in a random selection of households.

ii) asexual parasite and gametocyte prevalence and density will be determined by microscopic slide, rapid diagnostic test and molecular quantitative nucleic acid sequence based amplification (QT-NASBA) during cross-sectional surveys. Serum will also be collected for future analyses on malaria antibodies.

iii) the entomologic inoculation rate will be determined by mosquito catches by CDC light-trap in a random selection of houses in each cluster.

v) the human infectious reservoir will be determined by offering venous blood samples (3mL) to locally reared Anopheles mosquitoes in an experimental set-up.

The safety of the intervention will be determined in a selection of children 1 week after drug administration. Safety evaluation will concentrate on possible hemolysis, as assessed by haemoglobin concentration measured by hemocue and haptoglobin concentrations determined in serum.

ELIGIBILITY:
Inclusion Criteria:

* permanent resident of the research area
* age >1 years

Exclusion Criteria:

* severe anemia
* pregnancy

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
malaria morbidity by active and passive case detection. | during the entire study period
asexual parasite prevalence and density by microscopy, rapid diagnostic test and molecular QT-NASBA | monthly during the entire study period
gametocyte prevalence and density by QT-NASBA and microscopy | monthly during the entire study period
transmission intensity quantified by entomologic inoculation rate | continuously during the study period
human infectious reservoir | prior to the intervention and several months after the intervention

SECONDARY OUTCOMES:
asexual parasite and gametocyte density by microscopy and molecular QT-NASBA | monthly during the study period
human immune responses to malaria antigens | prior to the intervention and several months after the intervention
the prevalence of drug resistant parasite strains | prior to the intervention and several months after the intervention
Possible side effects of intervention with primaquine, notably hemolysis | one week after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Seif Shekalaghe, MPH MD, Principal Investigator — Kilimanjaro Christian Medical Centre; Robert Sauerwein, Prof MD PhD, Study Chair — Radboud University Medical Center; Frank Mosha, PhD, Study Director — Kilimanjaro Christian Medical Centre
Locations (1):
- Kilimanjaro Christian Medical Centre, Moshi, Tanzania

REFERENCES:
- [Background] von Seidlein L, Walraven G, Milligan PJ, Alexander N, Manneh F, Deen JL, Coleman R, Jawara M, Lindsay SW, Drakeley C, De Martin S, Olliaro P, Bennett S, Schim van der Loeff M, Okunoye K, Targett GA, McAdam KP, Doherty JF, Greenwood BM, Pinder M. The effect of mass administration of sulfadoxine-pyrimethamine combined with artesunate on malaria incidence: a double-blind, community-randomized, placebo-controlled trial in The Gambia. Trans R Soc Trop Med Hyg. 2003 Mar-Apr;97(2):217-25. doi: 10.1016/s0035-9203(03)90125-8. PMID 14584381
- [Background] Weerasinghe KL, Galappaththy G, Fernando WP, Wickremasinghe DR, Faizal HM, Wickremasinghe AR. A safety and efficacy trial of artesunate, sulphadoxine-pyrimethamine and primaquine in P falciparum malaria. Ceylon Med J. 2002 Sep;47(3):83-5. doi: 10.4038/cmj.v47i3.3434. PMID 12449772
- [Derived] Shah MP, Hwang J, Choi L, Lindblade KA, Kachur SP, Desai M. Mass drug administration for malaria. Cochrane Database Syst Rev. 2021 Sep 29;9(9):CD008846. doi: 10.1002/14651858.CD008846.pub3. PMID 34585740
- [Derived] Shekalaghe SA, Drakeley C, van den Bosch S, ter Braak R, van den Bijllaardt W, Mwanziva C, Semvua S, Masokoto A, Mosha F, Teelen K, Hermsen R, Okell L, Gosling R, Sauerwein R, Bousema T. A cluster-randomized trial of mass drug administration with a gametocytocidal drug combination to interrupt malaria transmission in a low endemic area in Tanzania. Malar J. 2011 Aug 24;10:247. doi: 10.1186/1475-2875-10-247. PMID 21864343
- [Derived] Shekalaghe SA, ter Braak R, Daou M, Kavishe R, van den Bijllaardt W, van den Bosch S, Koenderink JB, Luty AJ, Whitty CJ, Drakeley C, Sauerwein RW, Bousema T. In Tanzania, hemolysis after a single dose of primaquine coadministered with an artemisinin is not restricted to glucose-6-phosphate dehydrogenase-deficient (G6PD A-) individuals. Antimicrob Agents Chemother. 2010 May;54(5):1762-8. doi: 10.1128/AAC.01135-09. Epub 2010 Mar 1. PMID 20194698